CLINICAL TRIAL: NCT01322360
Title: A Multicenter, Open Label, Safety and Pharmacokinetic Study of Oral Morphine Sulfate Administration in Pediatric Subjects 2 Years Old Through 17 Years Old With Postoperative Pain
Brief Title: Safety and Pharmacokinetic Study of Oral Morphine Sulfate in Pediatric Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORP-OS+T-(2-17)-SPK-1
Record Dates: First submitted 2011-03-21; First posted 2011-03-24 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Morphine Sulfate (Other): oral solution (10 mg/5 mL or 20 mg/5 mL) or tablets (15 mg or 30 mg)given based on based on the current pediatric prescribing guidelines
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate
  Other Names: Morphine Sulfate Oral Solution; Morphine Sulfate Tablet

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of oral morphine sulfate in the treatment of postoperative pain in different pediatric age groups following multiple-dose administration.

To determine multiple-dose pharmacokinetics (PK) of morphine sulfate in pediatric subjects.

To compare plasma concentration of morphine sulfate in each age group of pediatric subjects with adult plasma morphine sulfate concentrations.

ELIGIBILITY:
Inclusion Criteria:

* parent or guardian provided written parental permission/informed consent, with subject assent (if required by local IRB).
* The child is 2 years old through 17 years old, inclusive (at the time of informed consent signing).
* A routine pediatric procedure is expected to require inpatient hospitalization postoperatively.
* Must be an inpatient for the study treatment period.
* Is expected by the investigator to require use of oral opioid for the treatment of postoperative pain.
* Has the ability to read and understand the study procedures and has the ability to communicate meaningfully with the study investigator and staff (if the subject is of preverbal age or cannot read or communicate meaningfully, then the subject's parent or guardian must meet this criterion).
* Child is expected to experience moderate to severe postoperative pain, in the investigator's opinion, during the immediate postoperative period after discontinuation of intermittent administration of IV opioid (preferably morphine) and is able to tolerate oral medications.
* If female subject is of childbearing potential, she must have a negative pregnancy test result at screening (serum) and on the day of surgery prior to surgery (urine).
* Must have vascular access to facilitate blood draws.

Exclusion Criteria:

* Has significant medical disease(s), laboratory abnormalities, or conditions(s) that in the investigator's judgment could compromise the subject's welfare, ability to communicate with study staff, complete study activities, or would otherwise contraindicate study participation. There is no minimum value for SpO2 for inclusion in the study; this should be based on the investigator's judgment.
* Has used opioids chronically (e.g., codeine, morphine, oxycodone, or hydromorphone, for >7 calendar days) within the previous 30 days.
* Has known hypersensitivity or contraindication to receiving oral opioid(s).
* Has a current active enteral malabsorption disorder.
* Has impaired liver function (e.g., alanine aminotransferase [ALT] ≥3 times the upper limit of normal [ULN], or bilirubin ≥3 times ULN), known active hepatic disease (e.g., hepatitis), evidence of clinically significant chronic liver disease or other condition affecting the liver (e.g., chronic hepatitis) that may suggest the potential for an increased susceptibility to hepatic toxicity with oral morphine exposure. Subjects with no previous history of liver function impairment may be enrolled prior to receipt of screening laboratory testing results.
* Has significantly impaired renal function or disease, as evidenced by an estimated glomerular filtration rate (i.e., from creatinine levels using the Schwartz formula) calculated to be less than one-third of normal for the applicable age of this study population. Subjects with no previous history of kidney function impairment may be enrolled prior to receipt of screening laboratory testing results.
* Has a history of substance abuse or there is evidence of current substance abuse, in the investigator's opinion.
* Has received epidural or regional anesthesia within 12 hours prior to the first dose of oral morphine sulfate.
* Has participated in an interventional clinical study (investigational or marketed product) within 30 days before screening, or plans to participate in another clinical trial in the next 30 days.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dante Landucci, M.D., Study Director — Quintiles, Inc.
Locations (11):
- United States (11):
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University Medical Center, Stanford, California
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital Medical Center of Akron d/b/a Akron Children's Hospital, Akron, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center of Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 06 May 2011 to 10 April 2012. A total of 75 subjects were screened and 50 subjects were enrolled (i.e., received at least 1 dose of study drug)
Pre-assignment Details: Only eligible pediatric subjects who signed the informed consent and completed all screening procedures within 14 days before the surgery were enrolled in the study.
Groups:
- Morphine Sulfate: Morphine sulfate oral solution and Morphine sulfate tablets
Period: Overall Study
Arm/Group | Morphine Sulfate
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Morphine Sulfate
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Adverse Events That Led to Study Discontinuation
Description: The primary safety endpoints were the percentage of subjects who experienced any AEs that led to study discontinuation, percentage of subjects with SAEs and those with a sedation score of 4. Secondary safety endpoints included the percentage of subjects who experienced any AEs of special interest, which included sedation, respiratory depression, nausea, vomiting, and pruritus of moderate to severe intensity/grade.
  Additional secondary endpoints were the incidence, type, relationship to study drug, and severity of AEs, and the percentage of subjects with clinically significant decreases in SpO2 and respiratory rate, as assessed by the investigator.
Time Frame: Up to 21 days
Population: 75 subjects were screened and 50 subjects took at least one dose of oral morphine sulfate.
Measure: Number; unit: participants
Groups:
- Morphine Sulfate: Subjects received morphine sulfate either as oral solution or tablet.
Arm/Group | Morphine Sulfate
Number analyzed (Participants) | 50
participants | 1

2. Secondary Outcome: Number of Subjects Who Experienced Adverse Events of Moderate to Severe Intensity / Grade
Description: Subjects who experienced any AEs of special interest, which included sedation, respiratory depression, nausea, vomiting, and pruritus of moderate to severe intensity/grade
Time Frame: Up to 21 days
Measure: Number; unit: participants
Groups:
- Morphine Sulfate: oral solution (10 mg/5 mL or 20 mg/5 mL) or tablets (15 mg or 30 mg)given based on based on the current pediatric prescribing guidelines
  Morphine Sulfate
Arm/Group | Morphine Sulfate
Number analyzed (Participants) | 50
participants | 19

ADVERSE EVENTS:
Time Frame: Adverse event reports began with first dose of study drug through end of study.
Arm/Group | Morphine Sulfate
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 35/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Sulfate (N=50)
Ileus (Gastrointestinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Sulfate (N=50)
Nausea (Gastrointestinal disorders) | 18 (18)
Constipation (Gastrointestinal disorders) | 17 (17)
Oxygen Saturation Decreased (Investigations) | 11 (11)
Pyrexia (General disorders) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Anxiety (Psychiatric disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days